CLINICAL TRIAL: NCT00727337
Title: Supplementing Hearing Aids With Computerized Auditory Training
Acronym: LACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C6303-R
Record Dates: First submitted 2008-07-30; First posted 2008-08-04 (Estimated); Results first posted 2015-01-13 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-06

CONDITIONS: Hearing Loss
Keywords: auditory perception; rehabilitation of hearing impaired
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- LACE-DVD (Experimental): Participants will complete the LACE training, however, not in an interactive computer mode but through a static DVD mode
  Interventions: Behavioral: Lace-DVD
- LACE-COMPUTER (Experimental): Participants will complete a computer-based auditory training program (i.e., LACE)
  Interventions: Behavioral: LACE-computer
- PLACEBO-DIRECTED LISTENING (Active Comparator): Participants will complete a directed listening to books on CD treatment
  Interventions: Behavioral: PLACEBO-Directed listening
- CONTROL (Active Comparator): Participants will be provided with hearing aids
  Interventions: Behavioral: CONTROL

INTERVENTIONS:
Behavioral: LACE-computer — Computerized Auditory Training
  Arms: LACE-COMPUTER
Behavioral: PLACEBO-Directed listening — Subjects will be asked to listen to books on tape for 20 minutes a day and answer questions as they go along
  Arms: PLACEBO-DIRECTED LISTENING
Behavioral: CONTROL — No specialized treatment will be provided in addition to standard of care audiology treatment provided with the provision of hearing aids
  Arms: CONTROL
Behavioral: Lace-DVD — DVD based Auditory Training
  Arms: LACE-DVD

SUMMARY:
The study is designed to examine the effectiveness of a computer-based auditory training program to improve the benefits received by individuals who wear hearing aids. The study will involve 3 groups - a computer-based training group, an active listening group which will involve listening to books on CD, and a placebo group that receives no additional treatment.

DETAILED DESCRIPTION:
This proposed study is a multi-site, single-masked (blinded), randomized controlled, parallel group clinical trial to assess the effectiveness of an at home PC-based auditory training as a supplement to standard-of-care hearing-aid intervention in veterans treated for hearing loss, with or without previous hearing-aid experience. The participants will be assigned randomly to one of three groups, with hearing-aid use stratified within the groups: (1) Group 1, HA+AT, in which the participants will receive standard-of-care hearing-aid intervention (HA) and complete the four-week LACE auditory training program (AT); (2) Group 2, HA, with the participants receiving only standard-of-care hearing-aid intervention (HA); and (3) Group 3, HA+DL, in which the participants will receive standard-of-care hearing-aid intervention (HA) and complete four-weeks of placebo auditory training, consisting of directed listening (DL) to books-on-tape. The participants in each group will attend four test sessions. During Session 1 the informed consent process will be completed, baseline assessments will be made to ensure that the participants meet the study inclusion criteria (page 52), testing of predictor variables (page 57-58) will be completed, and all hearing aids will be assessed for correct functionality (page 53). The participants then will be assigned randomly to a study group. Session 2 will occur four weeks after Session 1. During Session 2, baseline performance on the outcome measures will be assessed (page 54-57), as will performance on the predictor variables. Following testing, the participants in Groups 1 and 3 will receive training in the use of the AT or DL programs. Session 3 will occur at the end of the 4-week experimental training period. During Session 3 all participants will be retested on the outcome measures to assess short-term intervention outcomes. During Session 4, which will occur at seven-months post-study enrollment (i.e., six-months post training completion for Groups 1 and 3), all participants will be retested on all outcome measures to examine the long-term outcomes. In Sessions 2-4, the stability of hearing-aid function will be assessed through electroacoustic measures.

ELIGIBILITY:
Inclusion Criteria:

1. adult onset hearing loss,
2. English as the first language,
3. bilateral, symmetric, sensorineural hearing loss,
4. average audiometric thresholds for 500, 1000, and 2000 Hz less than 50-dB HL in either ear,
5. aided speech recognition in quiet of 40% binaurally,
6. appropriate cognitive skills assessed using the Mini Mental State Exam (Folstein et al., 1975) with age/education norms (Crum et al., 1993),
7. adequate vision to participate in the study as determined with the Smith-Kettlewell Institute Low Luminance (SKILL) Card,
8. eligible for VA-issued hearing aids.

Exclusion Criteria:

known neurological, psychiatric disorders, or co-morbid diseases that would prevent completion of the study as determined by chart review,

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2009-01; Primary Completion 2011-04 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Chisolm, PhD, Principal Investigator — University of South Florida
Locations (1):
- VA Medical Center, Bay Pines, Bay Pines, Florida, United States

REFERENCES:
- [Background] Chisolm TH, Saunders GH, Frederick MT, McArdle RA, Smith SL, Wilson RH. Learning to listen again: the role of compliance in auditory training for adults with hearing loss. Am J Audiol. 2013 Dec;22(2):339-42. doi: 10.1044/1059-0889(2013/12-0081). PMID 24018575
- [Result] Saunders GH, Smith SL, Chisolm TH, Frederick MT, McArdle RA, Wilson RH. A Randomized Control Trial: Supplementing Hearing Aid Use with Listening and Communication Enhancement (LACE) Auditory Training. Ear Hear. 2016 Jul-Aug;37(4):381-96. doi: 10.1097/AUD.0000000000000283. PMID 26901263

RESULTS

PARTICIPANT FLOW:
Groups:
- LACE-DVD: DVD-based auditory training
  Auditory Training with DVD: DVD based Auditory Training
- LACE - COMPUTER: Computer-based auditory training
  LACE: Computerized Auditory Training
- PLACEBO-DIRECTED LISTENING: Directed listening to books on CD
  Directed listening: Subjects will be asked to listen to books on tape for 20 minutes a day and answer questions as they go along
- CONTROL: No specialized treatment will be provided in addition to standard of care audiology treatment provided with the provision of hearing aids
  Usual care: No specialized treatment will be provided in addition to standard of care audiology treatment provided with the provision of hearing aids
Period: Overall Study
Arm/Group | LACE-DVD | LACE - COMPUTER | PLACEBO-DIRECTED LISTENING | CONTROL
Started | 68 | 65 | 73 | 73
Completed | 61 | 55 | 63 | 64
Not Completed | 7 | 10 | 10 | 9

BASELINE CHARACTERISTICS:
Groups:
- LACE-COMPUTER: Computer-based auditory training
  LACE: Computerized Auditory Training
- Total: Total of all reporting groups
Arm/Group | LACE-DVD | LACE-COMPUTER | PLACEBO-DIRECTED LISTENING | CONTROL | Total
Number analyzed (Participants) | 68 | 65 | 73 | 73 | 279
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 28 | 23 | 37 | 21 | 109
  >=65 years | 40 | 42 | 36 | 52 | 170
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (7.7) | 69 (7.8) | 67.1 (7.7) | 70 (7.3) | 68.6 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 68 | 65 | 73 | 73 | 279
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 68 | 65 | 73 | 73 | 279

OUTCOME MEASURES:

1. Primary Outcome: Words-in-Noise Test (WIN) Change
Description: Monosyllabic words (NU-6 female version) with a carrier phrase were presented auditory only in a multitalker babble.The participant is asked to repeat the last word of each phrase. The total number of correct words is input into the Spearman-Karber equation to derive a 50% point. This is the signal-to-noise ratio in dB that an individual requires to get 50% of the words correct. This test was completed at baseline and follow up visits.
Time Frame: Baseline, immediate post-intervention (up to 2 to 6 weeks), 6 month follow up
Population: Through the duration of the study, a total of 7 participants withdrew from LACE-DVD, 10 participants withdrew from LACE-C, 10 participants withdrew from Placebo, and 9 withdrew from the Control.
Measure: Mean (Standard Deviation); unit: dB SNR
Arm/Group | LACE-DVD | LACE-COMPUTER | PLACEBO-DIRECTED LISTENING | CONTROL
Number analyzed (Participants) | 68 | 65 | 73 | 73
dB SNR
  BASELINE | 9.8 (2.2) | 9.9 (2.7) | 9.7 (2.4) | 10.4 (2.3)
  POST-INTERVENTION: number analyzed (Participants) | 63 | 61 | 69 | 70
  POST-INTERVENTION | 9 (2.3) | 9.2 (2.7) | 9 (2) | 10 (2.3)
  6 MONTH FOLLOW UP: number analyzed (Participants) | 61 | 55 | 63 | 64
  6 MONTH FOLLOW UP | 9.3 (2.2) | 9.5 (2.4) | 9.4 (2.3) | 9.8 (2.2)

2. Secondary Outcome: Abbreviated Profile of Hearing Aid Benefit (APHAB) Change
Description: The Abbreviated Profile of Hearing Aid Performance (APHAP; Cox & Alexander 1995) was used to assess activity limitations and the Hearing Handicap Inventory for the Elderly or Adults (HHI; Ventry & Weinstein 1982; Newman et al. 1990) was used to assess participation restrictions. The APHAP is a 24-item questionnaire that documents hearing difficulties in specified listening situations. The items are answered on a 7-point scale from 'Always' (or 99%) to 'Never' (or 1%) with higher scores indicating greater reported hearing difficulty. The APHAP global score that ranges from 1 to 99 was used for all analyses.
Time Frame: Baseline, immediate post-intervention (up to 2 to 6 weeks), 6 month follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LACE-DVD | LACE-COMPUTER | PLACEBO-DIRECTED LISTENING | CONTROL
Number analyzed (Participants) | 68 | 65 | 73 | 73
units on a scale
  BASELINE | 32.3 (17) | 32 (18) | 34 (16) | 37 (18.2)
  POST-INTERVENTION: number analyzed (Participants) | 63 | 61 | 69 | 70
  POST-INTERVENTION | 31 (17) | 32 (16.55) | 32 (16) | 33.6 (16.1)
  6 MONTH FOLLOW UP: number analyzed (Participants) | 61 | 55 | 63 | 64
  6 MONTH FOLLOW UP | 30.45 (18.1) | 33.65 (17.75) | 33.15 (18.7) | 35.25 (16.45)

3. Secondary Outcome: Hearing Handicap Inventory for the Elderly (HHI) Change
Description: The HHI is a 25-item questionnaire that assesses the social and emotional consequences of hearing loss. The HHI for the elderly is for individuals age 65 years and older (Ventry & Weinstein 1982); the HHI for adults is for individuals aged 64 years and younger (Newman et al. 1990). The versions differ in the wording of three questions. The participants were asked to complete the appropriate HHI for aided listening to reflect their residual hearing handicap. HHI items are answered on a scale of Yes (4 points), Sometimes (2 points) and No (0 points), with higher scores indicating greater reported hearing handicap. Total HHI scores, which can range from 0 to 100, were used for all analyses.
Time Frame: Baseline, immediate post-intervention (up to 2 to 6 weeks), 6 month follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | LACE-DVD | LACE - COMPUTER | PLACEBO-DIRECTED LISTENING | CONTROL
Number analyzed (Participants) | 68 | 65 | 73 | 73
units on a scale
  BASELINE | 29.4 (22.6) | 31.3 (21.95) | 29.95 (20.15) | 33.8 (20.9)
  POST-INTERVENTION: number analyzed (Participants) | 63 | 61 | 69 | 70
  POST-INTERVENTION | 25.65 (19.65) | 29.35 (23.05) | 30.05 (19.3) | 29.35 (20.65)
  6 MONTH FOLLOW UP: number analyzed (Participants) | 61 | 55 | 63 | 64
  6 MONTH FOLLOW UP | 24.1 (19.7) | 27.85 (21.05) | 27.8 (19.55) | 32.45 (22)

ADVERSE EVENTS:
Arm/Group | LACE-DVD | LACE-COMPUTER | PLACEBO-DIRECTED LISTENING | CONTROL
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/65 | 0/73 | 0/73
Other Adverse Events (participants affected / at risk) | 0/68 | 0/65 | 0/73 | 0/73

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No